CLINICAL TRIAL: NCT04822272
Title: MagneThermoPro : Magnetic Resonance Thermography of Human Prostate
Acronym: ThermoPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2021/02
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer Diagnosis
Keywords: MRI; prostate; thermometry; laser; ablation

STUDY DESIGN:
Intervention Model Description: MRI sequence of 5 to 10 minutes to measure the variation of temprerature in the prostate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermometry MRI (Experimental): MRI sequence of 5 to 10 minutes to measure the variation of temprerature in the prostate
  Interventions: Device: MRI thermometry

INTERVENTIONS:
Device: MRI thermometry — MRI sequence of 5 to 10 minutes to measure the variation of temprerature in the prostate

SUMMARY:
The objective of this project is to offer a very innovative solution for measuring temperature variations in MRI on the prostate. Multiparametric prostate MRI can detect target lesions, on which targeted biopsies are then performed. The use of a temperature mapping on the prostate in MRI would make it possible to evaluate a focal treatment of the prostate by laser under MRI guidance

DETAILED DESCRIPTION:
Prostate MRI has become the benchmark examination to search for tumor targets, thanks to a multi-parameter protocol, including T2 sequences, diffusions, and T1 with gadolinium injection. A PIRADS prognostic score is performed on the different sequences and if the lesions are at high risk of malignancy (PIRADS 4 and 5), a targeted biopsy is performed. Minimally invasive ablations called focal treatments are developing more and more: HIFU, cryotherapy, laser, etc. Ultrasound remains the most widespread examination due to its availability, but with less sensitivity than MRI. Ablations are performed under ultrasound with fusion of MRI images In order to assess the ablation area under MRI, the measurement of temperature variations appears necessary to verify the effectiveness of ablation and the lesion volume. Temperature maps are feasible in cardiac MRI during radiofrequency. The thermal mapping MRI sequence is performed in cardiac MRI at the IHU in Bordeaux.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient with indication of injected multi-parameter MRI for the diagnosis of prostate cancer.
* Signed informed consent.
* Person affiliated or beneficiary of health insurance

Exclusion Criteria:

* MRI contraindications (Pace Maker, metallic foreign body, metallic heart valve).
* Contraindication to gadolinium salt,
* Patient under legal protection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
signal noise ratio | End of MRI exam (hour 1)
  the evaluation of the signal on the thermometry sequence

SECONDARY OUTCOMES:
temperature variance | End of MRI exam (hour 1)
  temperature variance measurements in a region of interest of the prostate
spatial distortion measurement | End of MRI exam (hour 1)
  spatial distortion measurement

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No